CLINICAL TRIAL: NCT00487617
Title: Endothelial Dysfunction Reversibility in Patients With Peripheral Arterial Disease
Brief Title: Arteriopathy and Endothelial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3801
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Arteriopathy; endothelial function; fruit juice
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fruit juice (Experimental): 300 mL of fruit juice
  Interventions: Procedure: Fruit juice or placebo absorption
- placebo (Placebo Comparator): 300 mL of fruit juice without polyphenols
  Interventions: Procedure: Fruit juice or placebo absorption

INTERVENTIONS:
Procedure: Fruit juice or placebo absorption — absorption of 300 ml of fruit juice ; 24 hours later, absorption of 300 ml of placebo.

SUMMARY:
To determine whether fruit juice might reverse endothelial dysfunction and whether this reversibility has a prognosis value

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arteriopathy
* Stable cardio-respiratory status

Exclusion Criteria:

* Dialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-10 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Endothelial function 1 hour after taking the juice | 1 hour after taking the juice

SECONDARY OUTCOMES:
Relationship between reversibility of the endothelial function and the patient's prognosis at 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rouyer, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service de Chirurgie Vasculaire, Strasbourg
  - Service de Physiologie et d'Explorations Fonctionnelles, Strasbourg